CLINICAL TRIAL: NCT06319820
Title: A Phase 3, Randomized Study Evaluating the Efficacy and Safety of TAR-210 Erdafitinib Intravesical Delivery System Versus Single Agent Intravesical Chemotherapy in Participants With Intermediate-risk Non-muscle Invasive Bladder Cancer (IR-NMIBC) and Susceptible FGFR Alterations
Brief Title: A Study to Evaluate TAR-210 Versus Single Agent Intravesical Cancer Treatment in Participants With Bladder Cancer
Acronym: MoonRISe-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 42756493BLC3004
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Non-Muscle Invasive Bladder Neoplasms
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — erdafitinib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Main Study: Group A: TAR-210 (Experimental): Participants in Group A will have TAR-210 inserted in the bladder on Day 1 and removed after 12 weeks. One TAR-210 will be inserted every 12 weeks over a treatment period of approximately 1 year.
  Interventions: Combination Product: TAR-210
- Main Study: Group B: MMC or Gemcitabine (Active Comparator): Participants in Group B will receive intravesical mitomycin C (MMC) or gemcitabine (investigator's choice) once weekly for 4 to 6 induction doses followed by a maintenance phase for a minimum of 6 months and up to 1 year.
  Interventions: Drug: Gemcitabine; Drug: MMC
- Substudy: Group A: TAR-210 (Experimental): Participants in Group A will have TAR-210 inserted in the bladder on Day 1 and removed after 12 weeks. One TAR-210 will be inserted every 12 weeks over a treatment period of approximately 1 year.
  Interventions: Combination Product: TAR-210
- Substudy: Group B: MMC (Active Comparator): Participants in substudy Group B will receive intravesical MMC once weekly for 4 to 6 induction doses followed by a maintenance phase for a minimum of 6 months and up to 1 year.
  Interventions: Drug: MMC

INTERVENTIONS:
Combination Product: TAR-210 — TAR-210 will be administered intravesically.
  Other Names: JNJ-42756493
  Arms: Main Study: Group A: TAR-210; Substudy: Group A: TAR-210
Drug: Gemcitabine — Gemcitabine will be administered intravesically.
  Arms: Main Study: Group B: MMC or Gemcitabine
Drug: MMC — MMC will be administered intravesically.
  Arms: Main Study: Group B: MMC or Gemcitabine; Substudy: Group B: MMC

SUMMARY:
The main purpose of this study is to compare the disease-free survival between participants receiving treatment with TAR-210 versus investigator's choice of intravesical chemotherapy for treatment of intermediate-risk NMIBC.

ELIGIBILITY:
Inclusion Criteria:

* Main study only: Have a histologically confirmed diagnosis (within 90 days of randomization) of IR-NMIBC with at least one of the following criteria fulfilled: a. Ta low grade (LG)/ Grade 1 (G1): primary or recurrent, b. Ta LG/G2: primary or recurrent and c. Greater than or equal to (>=) 1 of the following risk factors: i. Multiple Ta LG tumors, ii. Solitary LG tumor >= 3 cm, iii. Early recurrence (less than [<] 1 year), iv. Frequent recurrence (greater than [>] 1 per year), v. Recurrence after prior adjuvant intravesical treatment (single perioperative dose of chemotherapy does not fulfill this risk factor)
* Substudy only: Have a histologically confirmed new diagnosis (within 90 days of randomization) of IR-NMIBC for whom MMC is deemed the therapy of choice according to local standard of care with at least 1 of the following criteria fulfilled: a. Ta LG/G1, b. Ta LG/G2, and >=1 of the following risk factors: i) Multiple Ta LG tumors, ii) Solitary LG tumor >=3 cm
* Have a susceptible fibroblast growth factor receptor (FGFR) mutation or fusion either by urine testing or tumor tissue testing (from TURBT tissue), as determined by central or local testing
* Participants must be willing to undergo all study procedures (e.g., multiple cystoscopies from Screening through the end of study and TURBT for assessment of recurrence/progression) and receive the assigned treatment, including intravesical chemotherapy if randomized into that arm.
* Visible papillary disease must be fully resected prior to randomization and absence of disease must be documented at Screening cystoscopy
* Can have a prior or concurrent second malignancy (other than the disease under study) which natural history or treatment is unlikely to interfere with any study endpoints of safety or the efficacy of the study treatment
* Have an Eastern Cooperative Oncology Group performance status of 0 to 2

Exclusion Criteria:

* Known allergies, hypersensitivity, or intolerance to any study component or its excipients, including: a. Erdafitinib excipients; b.TAR-210 drug delivery system constituent materials ; c. urinary placement catheter materials; d. MMC or chemically related drugs; e. Gemcitabine or chemically related drugs
* Presence of any bladder or urethral anatomic feature (that is, urethral stricture) that, in the opinion of the investigator, may prevent the safe insertion, indwelling use, removal of TAR-210 or passage of a urethral catheter for intravesical chemotherapy
* Polyuria with recorded 24-hour urine volumes > 4000 milliliters (mL)
* Current indwelling urinary catheters, however, intermittent catheterization is acceptable
* Had major surgery or had significant traumatic injury and/or not fully recovered within 4 weeks before first dose (TURBT is not considered major surgery)

Substudy:

- Previous diagnosis of histologically confirmed urothelial bladder carcinoma at any time prior to current qualifying diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 561 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2028-06-28 (Estimated); Study Completion 2028-06-28 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) | From randomization to the date of the first documented recurrence, disease progression or death (approximately 4 years and 2 months)
  DFS is measured as the time from randomization to the date of the first documented recurrence of Ta non-muscle invasive bladder cancer (NMIBC) of any grade, disease progression, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Time to next Treatment (TTNT) | From randomization to the date of first documented subsequent treatment (local, systemic, surgical, or interventional) for bladder cancer (approximately 4 years and 2 months)
  TTNT is measured as the time from randomization to the date of first documented subsequent treatment (local, systemic, surgical, or interventional) for bladder cancer.
High Grade Recurrence-free Survival (HG RFS) | From randomization to the date of first documented evidence of HG NMIBC or death (approximately 4 years and 2 months)
  HG RFS is measured as the time from randomization to the date of first documented evidence of HG NMIBC or death, whichever occurs first
Progression Free Survival (PFS) | From randomization to the date of first documented disease progression or death (approximately 4 years and 2 months)
  PFS is measured as the time from randomization to the date of first documented evidence of disease progression or death, whichever occurs first.
Number of Diagnostic and Therapeutic Invasive Urological Interventions after Study Treatment | From study treatment completion up to trial discontinuation (approximately 4 years and 2 months)
  Number of diagnostic and therapeutic invasive urological interventions after study treatment, that is, endoscopic procedures (e.g., cystoscopies, transurethral resection of bladder tumors (TURBTs), ureteroscopies, urethral interventions, urethral stricture/bladder neck incision), catheterization (intravesical, suprapubic), intravesical treatments, major surgeries (e.g., radical cystectomy, simple cystectomy, urethroplasty) will be reported.
Number of Participants With Adverse Events (Including Physical Examination, Vital Signs and Laboratory Abnormalities) | From first dose up to 30 days after last dose of study treatment (approximately 4 years and 2 months)
  An AE is any untoward medical occurrence in a participant participating in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product, that does not necessarily have a causal relationship with the treatment. AEs will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0. Severity of AEs has 5 grades based on CTCAE criteria: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening and Grade 5: Death. Number of participants with adverse events (including physical examination, vital signs and laboratory abnormalities) will be reported.
Overall Survival (OS) | From randomization to the date of death (approximately 4 years and 2 months)
  OS is defined as the time from randomization to the date of death from any cause.
European Organization for Research and Treatment of Cancer-Quality of Life Questionnaire Core-30 items (EORTC-QLQ-C30) Scores | Baseline, Weeks 6, 12, 24, 36, and 48
  EORTC QLQ-C30 is a core 30-item questionnaire for evaluating the health-related quality of life (HRQoL) of participants participating in cancer clinical studies. It incorporates 5 functional scales (physical, role, cognitive, emotional, and social functioning), 3 symptom scales (fatigue, pain, and nausea or vomiting), and a global health status or HRQoL scale. Ratings for each item range from 1 (not at all) to 4 (very much). Higher scores indicated greater severity.
European Organization for Research and Treatment of Cancer-Quality of Life Questionnaire for Non muscle Invasive Bladder Cancer (EORTC-QLQ-NMIBC24) Scores | Baseline, Weeks 6, 12, 24, 36, and 48
  EORTC QLQ-NMIBC24 is a 24-item questionnaire for evaluating the HRQoL of participants with non-muscle-invasive bladder cancer. The questionnaire is designed to supplement the QLQ C30 and incorporates 6 multi-item scales and 5 single items. Ratings for each item range from 1 (not at all) to 4 (very much). Higher scores indicated greater severity.
Percentage of Participants With Significant Change From Baseline in EORTC-QLQ-C30 Scores | Weeks 6, 12, 24, 36, and 48
  EORTC QLQ-C30 is a core 30-item questionnaire for evaluating the HRQoL of participants participating in cancer clinical studies. It incorporates 5 functional scales (physical, role, cognitive, emotional, and social functioning), 3 symptom scales (fatigue, pain, and nausea or vomiting), and a global health status or HRQoL scale. Ratings for each item range from 1 (not at all) to 4 (very much). Higher scores indicated greater severity.
Percentage of Participants With Significant Change From Baseline in EORTC-QLQ-NMIBC24 Scores | Weeks 6, 12, 24, 36, and 48
  EORTC QLQ-NMIBC24 is a 24-item questionnaire for evaluating the HRQoL of participants with non-muscle-invasive bladder cancer. The questionnaire is designed to supplement the QLQ C30 and incorporates 6 multi-item scales and 5 single items. Ratings for each item range from 1 (not at all) to 4 (very much). Higher scores indicated greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Enterprise Innovation Inc. Clinical Trial, Study Director — Johnson & Johnson Enterprise Innovation Inc.
Locations (193):
- United States (38):
  - Arkansas Urology, Little Rock, Arkansas
  - Genesis Research LLC, Los Alamitos, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Irvine Medical Center, Orange, California
  - Genesis Research, San Diego, California
  - Genesis Research LLC, Sherman Oaks, California
  - University of Colorado Cancer Center Anschultz Cancer Pavilion, Aurora, Colorado
  - Colorado Clinical Research, Lakewood, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - First Urology, Jeffersonville, Indiana
  - Wichita Urology Group, Wichita, Kansas
  - Ochsner Health System, New Orleans, Louisiana
  - Chesapeake Urology Research Associates, Hanover, Maryland
  - Brigham And Women's Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Comprehensive Urology, Royal Oak, Michigan
  - Mercy Research, St Louis, Missouri
  - Specialty Clinical Research of St Louis, St Louis, Missouri
  - The Urology Center, PC, Omaha, Nebraska
  - Cancer Institute Of New Jersey, New Brunswick, New Jersey
  - Integrated Medical Professionals, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Associated Medical Professionals of Ny, Syracuse, New York
  - SUNY Upstate Med Univ, Syracuse, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Keystone Urology Specialists, Lancaster, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - The Conrad Pearson Clinic, Germantown, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Urology Associates, Nashville, Tennessee
  - Urology Austin, Austin, Texas
  - Urology Clinics of North Texas, Dallas, Texas
  - UT Southwestern, Dallas, Texas
  - Houston Metro Urology, Houston, Texas
  - Spokane Urology, Spokane, Washington
- Argentina (6):
  - Hospital Sirio Libanes, Buenos Aires
  - Investigaciones Clinico Moleculares (ICM), CABA
  - Cemaic Centro Privado de Especialidades Medicas Ambulatorias e Investigacion Clinica, Córdoba
  - Centro Urologico Profesor Bengio, Córdoba
  - Hospital Privado de la Comunidad, Mar del Plata
  - Sanatorio de la Mujer, Rosario
- Austria (5):
  - Medizinische Universitaet Graz, Graz
  - Medizinische Universitat Innsbruck, Innsbruck
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Universitaetsklinikum Salzburg Landeskrankenhaus, Salzburg
  - Medical University Vienna MUV, Vienna
- Belgium (7):
  - Onze -Lieve-Vrouwziekenhuis, Aalst
  - AZ Sint-Jan, Bruges
  - UZ Antwerpen, Edegem
  - AZ Maria Middelares, Ghent
  - Universitair Ziekenhuis Gasthuisberg, Leuven
  - Vitaz, Sint-Niklaas
  - CHU UCL Namur - Site Godinne, Yvoir
- Brazil (11):
  - Fundacao Pio XII, Barretos
  - Universidade Estadual De Campinas, Campinas
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - HBA SA Assitencia Medica e Hospitalar, Salvador
  - Fundacao do ABC Centro Universitario FMABC, Santo André
  - Irmandade Da Santa Casa De Misericordia De Sao Paulo, São Paulo
  - Fundacao Faculdade de Medicina - Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - Real e Benemérita Associação Portuguesa de Beneficência, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
- China (17):
  - Beijing Friendship Hospital Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Hunan Cancer hospital, Changsha
  - The Third People's Hospital of Chengdu, Cheng Du Shi
  - West China School of Medicine/West China Hospital, Sichuan University, Cheng Du Shi
  - Chongqing Cancer Hospital, Chongqing
  - Fujian Medical University Union Hospital, Fuzhou
  - Sun Yat Sen University Cancer Center, Guangzhou
  - Nanjing Drum Tower Hospital, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - Huadong Hospital Affiliated to Fudan University, Shanghai
  - The Second Hospital Of Tianjin Medical University, Tianjin
  - Cancer Hospital of Xinjiang Medical University, Ürümqi
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Tongji Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
- Czechia (5):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni Thomayerova nemocnice, Prague
  - Fakultni nemocnice v Motole, Prague
- Denmark (5):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - Odense Universitetshospital, Odense
  - Zealand University Hospital, Roskilde
- France (11):
  - Hospital Center University De Lille, Lille
  - Polyclinique de Limoges - Francois Chenieux, Limoges
  - Hôpital Edouard Herriot, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hopital Saint Louis, Paris
  - CHU Pitie Salpetriere, Paris
  - APHP - Hopital Bichat - Claude Bernard, Paris
  - Clinique de la Croix du Sud, Quint-Fonsegrives
  - Chu Rennes Hopital Pontchaillou, Rennes
  - CHU Rangueil, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (11):
  - Charite - Universitaetsmedizin Berlin (CCM), Berlin
  - Stadtisches Klinikum Braunschweig gGmbH-Klinik fur Urologie und Uroonkologie, Braunschweig
  - Studienzentrum Bayenthal, Cologne
  - Urologische Gemeinschaftspraxis, Dresden
  - Universitaetsklinikum Frankfurt, Frankfurt am Main
  - Urologikum Hamburg MVZ - Germany, Hamburg
  - Marien hospital Herne, Herne
  - Universitatsklinikum Jena, Jena
  - Klinikum rechts der Isar an der Technischen Universitat Munchen, München
  - Klinikum St. Elisabeth Straubing GmbH, Straubing
  - Katharinenhospital Innere Medizin, Stuttgart
- Hong Kong (2):
  - Prince Of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Ireland (4):
  - Cork University Hospital, Cork
  - Mater Misericordiae University Hospital, Dublin
  - Mater Private Hospital, Dublin
  - Adelaide and Meath Hospital, Dublin
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Hadassah University Hospita Ein Kerem, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Ziv Medical Center, Safed
  - Sourasky Medical Center, Tel Aviv
- Italy (9):
  - Ospedale S. Donato Arezzo, USL 8 - U.O. Oncologia Medica, Arezzo
  - Cliniche Humanitas Gavazzeni, Bergamo
  - ASST Spedali Civili Brescia, Brescia
  - Ospedale San Raffaele, Milan
  - Istituto Dei Tumori Di Milano, Milan
  - Universita Campus Bio-Medico di Roma, Roma
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Istituto Clinico Humanitas, Rozzano
  - A.O.Citta della Salute e della Scienza di Torino, Torino
- Japan (11):
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki Shi
  - St Marianna University Hospital, Kawasaki Shi
  - Kobe City Medical Center General Hospital, Kobe
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Osaka International Cancer Institute, Osaka
  - Gunma Prefectural Cancer Center, Ōta-ku
  - Saitama Medical Center, Saitama
  - JRC Wakayama Medical Center, Wakayama
  - Yokohama Municipal Citizen's Hospital, Yokohama
  - Yokohama City University Medical Center, Yokohama
  - Yokosuka Kyosai Hospital, Yokosuka
- Poland (10):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - IN VIVO Sp. z o.o, Bydgoszcz
  - Centrum Onkologii im Prof F Lukaszczyka w Bydgoszczy, Bydgoszcz
  - Uniwersytecki Szpital Kliniczny nr 4, Lublin
  - Wojewodzki Szpital im Sw Ojca Pio w Przemyslu, Przemyśl
  - Szpital Wojewodzki Im Sw Lukasza Samodzielny Publiczny Zaklad Opieki Zdrowotnej W Tarnowie, Tarnów
  - Medicover Integrated Clinical Services Sp z o o, Torun
  - Mazowiecki Szpital Onkologiczny Sp z o o, Wieliszew
  - 4 Wojskowy Szpital Kliniczny Z Poliklinika Samodzielny Publiczny Zaklad Opieki Zdrowotnej We Wroclawiu, Wroclaw
  - Dolnoslaskie Centrum Onkologii Pulmonologii i Hematologii, Wroclaw
- South Korea (6):
  - Chungbuk National University Hospital, Chungcheongbuk Do
  - National Cancer Center, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Seoul National University Hospital, Seoul
- Spain (16):
  - Hosp Univ A Coruna, A Coruña
  - Hosp. Univ. de La Ribera, Alzira
  - Fund. Puigvert, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Puerta Del Mar, Cadiz
  - Hosp. Gral. Univ. de Castellon, Castellon
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Clinica Univ. de Navarra, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp Virgen de La Victoria, Málaga
  - Hosp. Univ. Central de Asturias, Oviedo
  - Hosp.Univ.Parc Tauli, Sabadell
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Clinico Univ. de Valencia, Valencia
- Turkey (Türkiye) (7):
  - Adana Baskent Practice and Research Hospital, Adana
  - Ankara University Medical Faculty, Ankara
  - Dr Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - T C Saglik Bakanlıgi Goztepe Prof Dr Suleyman Yalcın Sehir Hastanesi, Istanbul
  - Kartal Dr Lutfi Kirdar sehir Hastanesi, Istanbul
  - Dokuz Eylul University Medical Faculty, Izmir
- United Kingdom (7):
  - Southmead Hospital, Bristol
  - St Bartholomews Hospital, London
  - Charing Cross Hospital, London
  - Newcastle Freeman Hospital, Newcastle upon Tyne
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Southampton General Hospital, Southampton
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency